CLINICAL TRIAL: NCT05696210
Title: Evaluation of the 1-year Prognosis of Patients Under Veno-arterial Extracorporeal Membrane Oxygenation for Cardiogenic Shock With Blood Transfusion Requirement
Acronym: HemoECMO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Klein Thomas, Medical Doctor, Central Hospital, Nancy, France
Other Study IDs: 2022PI060
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Blood Cells Transfusion; Transfusion Related Complication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High transfusion rate group: patients requiring Veno-arterial extracorporeal membrane oxygenation for medical or post cardiotomy cardiogenic shock and with a blood transfusion rate greater than or equal to 7 red blood cells.
  Interventions: Other: Transfusion rate of red blood cells
- Low transfusion rate group: patients who required Veno-arterial extracorporeal membrane oxygenation for medical or post cardiotomy cardiogenic shock and with a blood transfusion rate strictly below 7 red blood cells.

INTERVENTIONS:
Other: Transfusion rate of red blood cells — Transfusion rate of red blood cells greater than 7
  Groups: High transfusion rate group

SUMMARY:
The primary objective of this work is to study the 1-year prognosis of patients who received Veno-arterial extracorporeal membrane oxygenation for cardiogenic shock with the need for blood transfusion. Secondary objectives are to determine whether the transfusion strategy used (liberal or restrictive) still has an impact on overall mortality. We will also determine the factors associated with overall in-hospital mortality and look at the impact of transfusion in relation to the risk of hemolysis on the consequences in the occurrence of long-term chronic renal failure.

DETAILED DESCRIPTION:
The study of the prognostic impact of blood transfusion at 1 year in patients assisted by Veno-arterial extracorporeal membrane oxygenation in the context of cardiogenic shock would provide objective answers and optimize the decision to set up this assistance with regard to the possible long-term consequences. This decision currently remains at the discretion of the expert teams managing these patients.

The inclusion of patients in a state of cardiogenic shock under Veno-arterial extracorporeal membrane oxygenation with the need for transfusion, will therefore allow the elaboration of a multicentric observational study interested in the prognosis at 1 year of patients under VA ECMO according to the adopted transfusion threshold.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (> 18 years) at the time of data collection.
* Hospitalization in intensive care unit
* Cardiogenic shock of medical or surgical etiology according to the SCAI definition (stage B to E)
* Need for cardio-circulatory assistance such as Veno-arterial extracorporeal membrane oxygenation for at least 24 hours

Exclusion Criteria:

* - Age < 18 years
* In-hospital and out-of-hospital cardiac arrest.
* Veno-arterial extracorporeal membrane oxygenation set up at a center other than the study centers.
* Veno-arterial extracorporeal membrane oxygenation set up for less than 24 hours
* Death within 24 hours

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who were hospitalized between 2016 and 2021 for cardiogenic shock requiring Veno-arterial extracorporeal membrane oxygenation, outside the context of cardiac arrest, managed in the ICU.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2023-01-21 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
1-year survival | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 1 year
  To evaluate the association of blood transfusion (and its volume of administration) with the 1-year prognosis of patients managed with Veno-arterial extracorporeal membrane oxygenation for medical or post cardiotomy cardiogenic shock

SECONDARY OUTCOMES:
All-cause mortality rate during hospitalization for cardiogenic shock with the need for Veno-arterial extracorporeal membrane oxygenation | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  Assess the association between transfusion strategy as assessed by hemoglobin nadir during hospitalization with all-cause mortality.
30-day mortality | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 30 days
  To evaluate the association of blood transfusion (and its volume of administration) with the 30-day prognosis of patients managed with Veno-arterial extracorporeal membrane oxygenation for medical or postcardiotomy cardiogenic shock
Number of patients with stage 4 chronic kidney disease (GFR <30 mL/min) or with the need for chronic dialysis at 30 days. | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 30 days
  Assess the association of transfusion strategy with the occurrence of chronic renal failure (GFR <30 mL/min or with the need for chronic dialysis) at 30 days.
Number of patients with stage 4 chronic kidney disease (GFR <30 mL/min) or with need for chronic dialysis at 1 year. | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 1 year
  Evaluate the association of transfusion strategy with the occurrence of chronic renal failure (GFR <30 mL/min or with the need for chronic dialysis) at 1 year

REFERENCES:
- [Derived] Brouland M, Kimmoun A, Delmas C, Duarte K, Girerd N, Vardon-Bounes F, Klein T. Association Between Red Blood Cells Transfusion and 1 Year Mortality in Patients on Venoarterial Extracorporeal Membrane Oxygenation for Cardiogenic Shock. ASAIO J. 2025 Oct 1;71(10):833-840. doi: 10.1097/MAT.0000000000002424. Epub 2025 Apr 2. PMID 40171953